CLINICAL TRIAL: NCT05305859
Title: A Multi-center, Prospective, Single-arm Study of Venetoclax Combining Chidamide and Azacitidine (VCA) in the Treatment of Refractory/Relapsed Acute Myelogenous Leukemia (R/R AML)
Brief Title: Venetoclax Combining Chidamide and Azacitidine (VCA) in the Treatment of R/R AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Collaborators: Fujian Provincial Hospital (Other); Fujian Cancer Hospital (Other Government); Zhangzhou manicipal hospital of Fujian Province (Unknown); Jieyang People's Hospital (Other); Dongguan People's Hospital (Other Government); Huizhou Municipal Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FXMH-AML-001; ChiCTR2200056657 (Registry Identifier: Chinese clinical trial registry)
Record Dates: First submitted 2022-03-08; First posted 2022-03-31 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Leukemia, Myeloid, Acute; Relapsed Adult AML; Refractory Leukemia
Keywords: refractory/relapsed acute myelogenous leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- venetoclax combining chidamide and azacitidine (VCA) (Experimental): 28 days per cycle × at least 2 cycles；
  1) chidamide 30mg biw × 2weeks；2) venetoclax 200mg/d × 2 weeks 3) azacitidine 100mg/d d1-7
  Interventions: Drug: venetoclax combining chidamide and azacitidine (VCA)

INTERVENTIONS:
Drug: venetoclax combining chidamide and azacitidine (VCA) — information already included in arm/group descriptions
  Other Names: VCA

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Venetoclax Combining Chidamide and Azacitidine (VCA) in the Treatment of relapsed and/or refractory AML

DETAILED DESCRIPTION:
Patients with relapsed and/or refractory AML have inferior outcomes. The regimen of Venetoclax and Azacitidine has been widely used in the treatment of RR AML and has proved to achieve CR rate of 30% ~ 40%. However, the median duration of response (DOR) of this regimen is about one year. Chidamide is a histone deacetylase (HDAC) inhibitor and preclinical data showed adding low-dose Chidamide to venetoclax could significantly promoted apoptosis of leukemia cell lines. Meanwhile, the Venetoclax Combining Chidamide and Azacitidine (VCA) regimen was applied to 2 patients with refractory AML. This regimen was well tolerated and both patients achieved CR after one cycle. Thus, we register this clinical trial and evaluate the safety and efficacy of VCA regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Relapsed and refractory patients with acute myeloid leukemia via morphology and immunology
* ECOG：0-2
* Life expectancy ≥ 3 months
* Adequate laboratory parameters during the screening period as evidenced by the following:

  1. Creatinine clearance≥30 mL/min and serum Creatinine ≤ 160µmol/L
  2. ALT and AST ≤ 3 × upper limit of normal (ULN)
  3. Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL)
* Central nervous system leukemia
* Uncontrolled or significant cardiovascular disease, including any of the following:

  1. Bradycardia of less than 50 beats per minute, unless the subject has a pacemaker; Diagnosis of or suspicion of long QT syndrome (including family history of long QT syndrome);
  2. Systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg; History of clinically relevant ventricular arrhythmias (eg, ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes);
  3. History of second (Mobitz II) or third degree heart block (subjects with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker);
  4. History of uncontrolled angina pectoris or myocardial infarction within 6 months prior to Screening;
  5. History of New York Heart Association Class 3 or 4 heart failure;
  6. Complete left bundle branch block;
  7. Known history of left ventricular ejection fraction (LVEF) ≤45% or less than the institutional lower limit of normal;
* Active acute or chronic systemic fungal, bacterial, or viral infection not well controlled by antifungal, antibacterial or antiviral therapy;
* Suffered from other non-myeloid malignancies within 2 years, except adequately treated non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated with no evidence of disease
* Females who are pregnant or breastfeeding;
* Mental disorders that hinder research participation
* Previous solid organ transplantation (SCT treatment is allowed in advance, but if the patient has GVHD or is still receiving immunosuppression/GVHD treatment, it is not allowed)
* Any other situation where the investigator believes that the patient should not participate in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) rate | 2 months
  CR was <5% marrow blasts by morphology
Overall response rate (ORR) | 2 months
  ORR is defined as CR, CRi and PR.

SECONDARY OUTCOMES:
1 year leukemia free survival (LFS) | 1 year from treatment initiation
  Leukemia-free survival (LFS) is defined as survival without evidence of relapse from treatment initiation
1year overall survival (OS) | 1 year from treatment initiation
  Overall survival（OS）is defined as the time from treatment initiation to death from any cause.
Adverse events | 2 months
  Adverse event is defined as any untoward medical occurrence associated with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, Principal Investigator — The First Affiliated Hospital of Xiamen University
Locations (1):
- Bing Xu, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No